CLINICAL TRIAL: NCT06453382
Title: Development and Testing of a Sub-district Specific Model of 'Whole-of-government', and 'Whole-of-society' Approaches for the Prevention and Control of Non-communicable Diseases in a Sub-district of Bangladesh
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BRAC University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-10 November'22-045
Record Dates: First submitted 2024-05-14; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; Diabetes; Asthma; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Non-communicable disease; Hypertension; Diabetes; Chronic respiratory disease; Whole of government; Whole of society
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Asthma; Pulmonary Disease, Chronic Obstructive; Noncommunicable Diseases | interventions — Mass Screening

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 'Whole of government' and 'whole of society' approach (Experimental): Sub-district level potential human resources engagement to control and prevent NCDs
  Interventions: Behavioral: Behavioural change modification, Screening, NCD related knowledge practice and attitude

INTERVENTIONS:
Behavioral: Behavioural change modification, Screening, NCD related knowledge practice and attitude — The investigators will provide periodic training regarding the control and prevention of NCDs to the stakeholders. The investigators will provide WHO-Package of Essential Non-Communicable Diseases (PEN) protocol training to the stakeholders involved in healthcare service delivery. The investigators will equip the government healthcare facilities with the equipment needed for the screening of NCDs. For the stakeholders who are not directly involved with healthcare service delivery, the investigators will train them about the 5 NCDs (diabetes, hypertension, chronic respiratory disease, cancer, and mental illness) and the 5 NCD risk factors (unhealthy diet, inadequate physical activity, tobacco cessation, alcohol cessation, and air pollution). The investigators will also share information, education, and communication (IEC) materials with the stakeholders, and then they will share the information with the community.

SUMMARY:
Globally, non-communicable diseases (NCDs) are the leading cause of both mortality and morbidity. This intervention study aims to prevent and manage NCDs by adopting the World Health Organization's (WHO) comprehensive 'whole-of-government' and 'whole-of-society' approach. Although the Bangladesh government has devised a Multisectoral Action Plan (MAP) for NCD prevention and control, there's a need to operationalize these approaches at the sub-district level. This requires establishing a framework, implementing it, and assessing its effectiveness. To accomplish the study's objectives, the investigators will initially identify key stakeholders involved in NCD-related work or potentially able to contribute. Subsequently, investigators will qualitatively explore their potential involvement in NCD prevention and control, including their current roles and responsibilities, and how they could further contribute. Workshops will be conducted with these stakeholders to develop a tailored intervention model for NCD prevention and control at the sub-district level, utilizing the 'whole-of-government' and 'whole-of-society' approach. Following this, the sub-district specific model will be implemented, and the process will be documented. Finally, an evaluation will be conducted to assess the effectiveness of the sub-district specific model in achieving NCD-specific outcomes.

DETAILED DESCRIPTION:
1. Aims:

   To generate evidence of 'whole-of-government' and 'whole-of-society' approach for non-communicable diseases (NCD) prevention and control in Bangladesh
2. General objective:

   The general objective of the research is to develop and test an sub-district-specific multi-sectoral model of 'whole-of-government' and 'whole-of-society' approach for NCD prevention and control in Birganj sub-district of Dinajpur district.
3. Specific Objectives:

   * Identify government, non-government (NGO), and civil-society organizations (CSO) relevant to the prevention and control of NCDs
   * Define the roles and responsibilities of the government, NGO, and CSOs pertinent to the prevention and control of NCDs
   * Develop an sub-district specific intervention model of 'whole-of-government' and 'whole-of-society' approach for NCD prevention and control
   * Implement the sub-district specific model and carry out a process documentation
   * Evaluate the sub-district specific model with regard to NCD specific outcomes
4. Rationale In 2018, the Government of Bangladesh launched a multisectoral action plan (MAP) in alignment with the World Health Organization (WHO) Global Action Plan for the prevention and control of NCD. The core elements of this MAP for prevention and control of NCD is 'whole-of-government' and 'whole-of-society' approach, universal health coverage, cultural relevance, reduction of inequity, and life-course approach. The MAP outlined four action areas: i. advocacy, leadership, and partnership, ii. health promotion and risk reduction, iii. health system strengthening for early detection and management of NCDs and their risk factors, and iv. surveillance, monitoring and evaluation, and research. The MAP also provides guidelines for multi-sectoral coordination mechanisms for the implementation of the action areas. In the MAP, the guidelines for the formulation of sub-district level multisectoral committee and functions of the committees have been described. However, to implement the 'whole-of-government' and the 'whole-of-society' approaches at the sub-district level, there is a need to develop a model, implement the model and evaluate the effectiveness of the model. Accordingly, in this study, the investigators propose developing a sub-district specific 'whole-of-government' and 'whole-of-society' model to prevent and control NCD and evaluate the model's effectiveness.
5. Methodology (Brief):

   As NCD is a broad area, investigators will follow the WHO 5 by 5 framework (five diseases and five risk factors) as a guide for implementing the research. Accordingly, the focus of our research will be five risk factors: i. Tobacco consumption, ii. Alcohol consumption, iii. Unhealthy diet, iv. Physical inactivity, and v. Air pollution, and five diseases: i. Cardiovascular diseases, ii. Diabetes, iii. Cancers, iv. Chronic respiratory diseases, and iv. Mental Health Disorders.

   The study will be implemented in Birganj, an sub-district of Dinajpur district. As per the 2011 census, Birganj sub-district has 317252 (159612 male and 157641 female) population. In the sub-district, firstly, the investigators will identify the current government, NGO, and CSOs and their possible roles for NCD prevention and control using a landscape analysis. In the second step, in collaboration with the Directorate General of Health Services, the investigators will define the NCD prevention and control roles and responsibilities of the identified organizations. In the third step, investigators will arrange workshops and meetings with the representatives from the organizations (government: local government and sub-district administration, health, police, education, women affairs, social affair, agriculture, fisheries, livestock, engineering; NGOs, and civil society organizations (CSOs) and develop an sub-district specific model of 'whole-of-government' and 'whole-of-society' approach for NCD prevention and control. In collaboration with the government, NGO and CSO, and under direction from the non-communicable diseases control (NCDC) of the Directorate General of Health Services (DGHS), the investigators will implement the model for one year and evaluate the effectiveness of the model on the indicators of both supply side, and demand side. On the supply side, investigators will evaluate whether the involved organizations developed an understanding of the whole-of-government' and 'whole-of-society' approach and the service delivery and readiness of each of them improved or not. On the demand side, the investigators will evaluate the changes in the NCD risk factors among the adults and the adolescents, changes in the adherence to medication and lifestyle measures among the people with NCDs, the changes in the proportion of population screened for the five NCDs, and five risk factors mentioned above, and the changes in the proportion of people with control over blood pressure, blood sugar, total cholesterol, and lungs function. In this research, the investigators will administer both qualitative and quantitative methodology. The evaluation of the model will be done primarily through quantitative methods using a pre-post design. There will be a process documentation component to document barriers and facilitators of the implementation so that this model can be scaled up in other settings.
6. Ethical clearance: Ethical clearance for this study will be obtained from the Institutional Review Board (IRB) of Bangladesh Rehabilitation Assistance Committee (BRAC) James P Grant School of Public Health, BRAC University. Informed written consent will be taken from each participant. Participation will be voluntary, and the participants will have the right to withdraw at any time of the study.
7. Impact of the study in future research: Through this research, the investigators will develop and test an sub-district specific model of 'whole-of-society' and 'whole-of-government' approach for prevention and control of NCD. If the model is successful, there will be further research on the improvement and scalability of the model.
8. Impact of the study at national level:

If the sub-district specific model of 'whole-of-society' and 'whole-of-government' approach for prevention and control developed and tested through this study shows results, the model can be scaled-up in other sub-districts of Bangladesh. In the long run, this research will help the government of Bangladesh achieve the NCD related targets of the multi-sectoral action plan, global action plan and the sustainable development goal (SDG) and relevant targets (Goal 3, target 3.4, 3.5, 3.6, 3.8, 3.9, 3.A, and 3.C)

ELIGIBILITY:
Inclusion Criteria:

* Work within the area of study site

Exclusion Criteria:

* Do not work within the area of study site

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of trained healthcare providers in government healthcare facility in sub-district changes | 2 years
  We will perform a baseline service availability and readiness assessment of the healthcare facility using a tool adapted from WHO's harmonized health facility assessment tool. After that, at the end line, we again perform service availability and readiness assessments of those particular healthcare facilities.
Number of equipment/logistics in government healthcare facility in sub-district changes | 2 years
  We will perform a baseline service availability and readiness assessment of the healthcare facility using a tool adapted from WHO's harmonized health facility assessment tool. After that, at the end line, we again perform service availability and readiness assessments of those particular healthcare facilities.
Change in the proportion of physical activity, tobacco consumption, fruits and vegetable consumption among adolescents and adults | 2 years
  We will conduct baseline and end line community survey of adolescent and adult participants. From there, we will measure the change of the proportions of the NCD risk factors.
Prevalence of NCDs reduced among the adults (>/= 18 years) | 2 years
  We will conduct baseline and end line community survey of adolescent and adult participants. From there, we will measure the change of the proportions of the NCD risk factors.
Proportion of adherence to medication and lifestyle modification measures change among the people with NCDs | 2 years
  We will conduct baseline and end line community survey of adolescent and adult participants. From there, we will measure the change of the proportions of the NCD risk factors.
The proportion of people with control of hypertension, lung function, and blood sugar increased | 2 years
  We will conduct baseline and end line community survey of adolescent and adult participants. From there, we will measure the change of the proportions of the NCD risk factors.
The proportion of adults screened for cancer, diabetes, mental health disorders, hypertension and chronic respiratory diseases increased | 2 years
  We will conduct baseline and end line community survey of adolescent and adult participants. From there, we will measure the change of the proportions of the NCD risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Malay K Mridha, PhD, Principal Investigator — BRAC James P Grant School of Public Health, BRAC University
Locations (1):
- BRAC James P Grant School of Public Health, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request to the central contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code